CLINICAL TRIAL: NCT00247156
Title: An Investigation Into the Effectiveness of NAET on Autism Spectrum Disorders
Brief Title: An Autism Study Using Nambudripad's Food Allergy Elimination Treatments
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nambudripad's Allergy Research Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: narfoundationautismstudy; narffoundation 101
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2006-04

CONDITIONS: Autism; Food Allergies
Keywords: Autism; eye contact; Noncommunicable
MeSH Terms: conditions — Autistic Disorder; Food Hypersensitivity

INTERVENTIONS:
Procedure: Acupressure treatments and NAET treatments

SUMMARY:
1. We hypothesize that children in the experimental group will show a significant improvement over the control group as all food allergens groups and some other relevant allergenic substances are desensitized in a systematic way using the NAET® methodology within the specified period of study.

DETAILED DESCRIPTION:
An autism Pilot Study Using NAET (Nambudripad's Allergy Elimination Techniques)

Aim/Question:

The principle goal of this proposed study (pilot study) is to test the efficacy of NAET® (Nambudripad's Allergy Elimination Technique) protocols for the treatment of Autism Spectrum Disorder in children between the ages of 3-10 years old, especially in the areas of improving language and communication skills.

To elaborate further, the NAET® protocols uses chiropractic/acupuncture manipulation of spinal nerve roots to alert the nervous system about the presence of the allergen in the hand and thus to wake up the dormant sensory nerve fibers (the sympathetic and parasympathetic nerve fibers) that carry messages from the periphery to the association cortex of the brain, through spinal nerves of the body, as well as from the brain to the periphery and target organs (also known as afferent and efferent nerves). This is followed by acupressure massage on specific acupuncture points to balance the energy of the entire nervous system. Avoidance of the treated allergen/substance for 24 hours after treatment completes the NAET® treatment protocol.

When we enroll them into NAET program, most of them are nonverbal and non-communicable. But by the time they complete 10 to 15 NAET basic treatments for an allergy to essential nutrients, most of them start verbal and nonverbal communications, social interactions, playing with other children, improve sleep, reduce restlessness, reduce irritability, reduce abnormal body movements like flapping hands, pulling hair, etc., and start behaving like normal children. When they finish the complete NAET program most of them become normal again.

The complete NAET program usually takes about 75-100 office visits over a span of couple of years.

Method:

The NAET® method has been highlighted in literature (Nambudripad DS: Say Goodbye to Illness, Third Edition, Delta Pub 1999, 136-137; Nambudripad DS: Say Good-bye to Allergy-related Autism. Delta Pub 2001; The Journal of NAET Energetics and complementary medicine 1 (1) 76-79, 2005, The Journal of NAET Energetics and complementary medicine 1 (1) 85-86, 2005, Tsering: Natural Health 29 (6) 80-85, 1999, and and Teuber and Porch-Curren: Curr Opin Allergy Clin Immunol 3:217-221, 2003).

NARF IRB Approval:

After the design and conceptualization of this clinical project, a summary of the project was submitted to the Nambudripad's Allergy Research Foundation Institutional Review Board. The NARF IRB will study the project and would meet to discuss the pros and cons of this project. There will be external physicians whose specialization would include pediatrics and child welfare to evaluate the project and the ethical treatment to children. (The board after asking several questions approved this study unanimously in October 2004. The Board also requested for periodic (every six months) updates on the progress of this project).

NAET ALLERGENS TO TREAT AUTISM

1. Egg Mix
2. Calcium mix
3. Vitamin C
4. B complex vitamins
5. Sugar Mix
6. Iron Mix
7. Vitamin A
8. Mineral Mix
9. Heavy Metals
10. Salt Mix
11. Corn Mix
12. Grain Mix
13. Artificial Sweeteners
14. Yeast Mix
15. Stomach acid
16. Digestive enzymes
17. Neurotransmitters
18. Immunizations and Vaccinations: either you received or your parent received before you were born. Test them individually and if found treat them individually.

    (MMR: (measles, mumps, rubella), DPT: (diphtheria, pertussis, tetanus), Polio vaccine, Small pox, Chickenpox, Influenza, hepatitis-B, hepatitis C.)
19. Pesticides
20. Alcohol
21. Coffee Mix
22. Nut Mix 1
23. Nut Mix 2
24. Spice Mix 1
25. Spice Mix 2
26. Animal Fats
27. Vegetable Fats
28. Vitamin F (
29. Dried Bean Mix
30. Amino Acids-1
31. Amino Acids 2
32. Dimethyl Glycine
33. Food additives
34. Food colors
35. Night-shade vegetables
36. Starch Complex
37. Drugs with allergy: Antibiotics (Individual antibiotics)
38. Hormones
39. Baking powder/ Baking soda
40. School work materials
41. Fabrics
42. Water
43. Chemicals
44. Plastics
45. Hypothalamus
46. Brain Tissue
47. Parts of the Brain
48. Other enzymes
49. Perfume mix
50. Tobacco smoke

ELIGIBILITY:
Inclusion Criteria:

Volunteers will be selected based on the well-defined inclusion criteria such as all control and sample children showed typical autistic symptoms before NAET® treatment: made no eye contact, unable to talk and communicate. All subjects (both control and sample) should be within the age limit of 3 to10 years and should have established and demonstrated autism spectrum disorder by a conventional physician. -

Exclusion Criteria:

Any child that has a history of various complications of illness other than autism spectrum disorder would be disqualified. Previously treated with NAET treatments for this condition will be disqualified to enroll in the study. Any patient who has any of the following incidents will also be disqualified.

1. Previous surgeries, congenital deformities of heart, lung, liver, brain, kidney, etc.
2. Any type of cancer
3. Aids
4. Any physically debilitating disorders and diagnosed mental retardation, Down's syndrome, etc.
5. Children with the history of severe allergies or anaphylactic reactions will be rejected.

   -

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2004-11; Study Completion 2005-11

PRIMARY OUTCOMES:
Improvement in speech and communication

SECONDARY OUTCOMES:
Elimination or reduction of commonly seen autistic traits

CONTACTS AND LOCATIONS:
Overall Officials: Devi S. Nambudripad, LAc, PhD, Principal Investigator — The journal of NAET Energetics and Complementary Medicine
Locations (1):
- PNIB Research Center, Buena Park, California, United States